CLINICAL TRIAL: NCT00694629
Title: TBTC Study 29: Evaluation of a Rifapentine-containing Regimen for Intensive Phase Treatment of Pulmonary Tuberculosis
Brief Title: TBTC Study 29: Rifapentine During Intensive Phase Tuberculosis (TB) Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-5399; NCT01043575 (obsolete NCT alias)
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Tuberculosis
Keywords: pulmonary tuberculosis; treatment
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; rifapentine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): rifampin, isoniazid, pyrazinamide, ethambutol
  Interventions: Drug: rifampin
- 2 (Experimental): rifapentine 10 mg/kg, isoniazid, pyrazinamide, ethambutol
  Interventions: Drug: rifapentine
- 3 (Experimental): rifapentine 15 mg/kg, isoniazid, pyrazinamide, ethambutol
  Interventions: Drug: rifapentine
- 4 (Experimental): rifapentine 20 mg/kg, isoniazid, pyrazinamide, ethambutol
  Interventions: Drug: rifapentine

INTERVENTIONS:
Drug: rifampin — tablet, 10 mg/kg, daily, 8 weeks
  Other Names: Rifadin
  Arms: 1
Drug: rifapentine — tablet, 10 mg/kg, daily, 8 weeks
  Other Names: Priftin
  Arms: 2
Drug: rifapentine — tablet, 15 mg/kg, daily, 8 weeks
  Other Names: Priftin
  Arms: 3
Drug: rifapentine — 20 mg/kg, daily, 8 weeks
  Other Names: Priftin
  Arms: 4

SUMMARY:
Protocol Synopsis The goal of this Phase 2 clinical trial is to evaluate the antimicrobial activity and safety of an experimental intensive phase (first 8 weeks of treatment) tuberculosis treatment regimen in which rifapentine is substituted for rifampin.

Primary Objective

* To compare the antimicrobial activity and safety of standard daily regimen comprised of rifampin (approximately 10 mg/kg/dose) + isoniazid + pyrazinamide + ethambutol (RHZE) to that of an experimental regimen comprised of rifapentine (approximately 10 mg/kg/dose) + isoniazid + pyrazinamide + ethambutol (PHZE).

Secondary Objectives

* To determine and compare for each regimen the time to culture-conversion, using data from 2-, 4-, 6-, and 8-week cultures (10, 20, 30, 40 doses).
* To determine and compare for each regimen the proportion of patients with any Grade 3 or 4 adverse reactions
* To determine the correlation of the MGIT/BACTEC liquid culture growth index and other mycobacterial and clinical biomarkers with time to culture conversion and treatment failure
* To store serum for future assessment of biomarkers of TB treatment response and hypersensitivity to study drugs.
* To compare adverse events and 2-month culture conversion rates among HIV-infected patients vs. HIV-uninfected patients
* To determine the tolerability and safety, and estimate the antimicrobial activity, of experimental regimens that include isoniazid + pyrazinamide + ethambutol plus either rifapentine 15 mg/kg/dose or rifapentine 20 mg/kg/dose, all administered daily. Assessment of these doses of rifapentine will be performed as an extension to the main study after enrollment in the main study has been completed.

Design

This will be a prospective, multicenter, open-label clinical study. Adults suspected of having pulmonary tuberculosis who meet eligibility criteria will be randomized to receive either the experimental intensive phase tuberculosis treatment regimen or the standard intensive phase tuberculosis treatment regimen. Randomization will be stratified by presence/absence of cavitation on baseline chest radiograph, and by geographic continent. All doses of study drugs will be given under direct observation and administered 5 days per week. After a subject completes intensive phase therapy, he/she then will be treated with a non-experimental continuation phase tuberculosis treatment regimen.

The study extension will be a prospective, multicenter clinical trial. Eligibility criteria will be the same as for the main study. Participants will be randomized to one of four regimens: the standard intensive phase treatment regimen, an investigational regimen in which rifapentine 10 mg/kg/dose is substituted for rifampin, an investigational regimen in which rifapentine 15 mg/kg/dose is substituted for rifampin, or an investigational regimen in which rifapentine 20 mg/kg is substituted for rifampin. Randomization will be stratified by the presence/absence of cavitation on baseline chest radiograph, and by study site. Study drugs will be administered 7 days per week. After a subject completes intensive phase therapy, he/she then will be treated with a non-experimental continuation phase tuberculosis treatment regimen. Subjects will have blood drawn for one pharmacokinetic determination of rifapentine concentration at or after the week 2 visit during intensive phase therapy.

This study is being conducted in 2 phases.

1. The main study compares a 10 mg/kg dose of rifapentine, open label, against 10 mg/kg rifampin in an otherwise standard intensive phase regimen of treatment for pulmonary tuberculosis. The projected sample size was 480 enrollments; 530 patients were actually enrolled.
2. The study extension evaluates higher doses of rifapentine, with the specific rifapentine doses (10 mg/kg, 15 mg/kg, and 20 mg/kg) blinded to patients and clinicians, with data collection and endpoints otherwise similar to the main study. The projected sample size for the study extension is 320 enrollments.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected pulmonary tuberculosis with acid-fast bacilli in a stained smear of expectorated or induced sputum.
2. Willingness to have HIV testing performed, if HIV serostatus is not known or if the last documented negative HIV test was more than 3 months prior to enrollment.
3. 5 (five) or fewer days of multidrug therapy for tuberculosis disease in the 6 months preceding initiation of study drugs.
4. 7 (seven) or fewer days of fluoroquinolone therapy in the 30 days preceding initiation of study drugs.
5. Age >= 18 years
6. Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs; see Appendix B)
7. Signed informed consent
8. Women of child-bearing potential must agree to practice an adequate (barrier) method of birth control or to abstain from heterosexual intercourse during study therapy.
9. Laboratory parameters done within 14 days prior to, enrollment:

   * Serum or plasma alanine aminotransferase (ALT) activity ≤ 3 times the upper limit of normal
   * Serum or plasma total bilirubin level ≤ 2.5 times the upper limit of normal
   * Serum or plasma creatinine level ≤ 2 times the upper limit of normal
   * Complete blood count with hemoglobin level of at least 7.0 g/dL
   * Complete blood count with platelet count of at least 100,000/mm3
   * Negative pregnancy test (women of childbearing potential)

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Known intolerance or allergy to any of the study drugs
3. Concomitant disorders or conditions for which isoniazid (INH), rifamycins, pyrazinamide (PZA), or ethambutol (EMB) are contraindicated. These include severe hepatic damage, acute liver disease of any cause, and acute uncontrolled gouty arthritis.
4. Current or planned therapy, during the intensive phase of TB therapy, with combination antiretroviral therapy for HIV, or with cyclosporine or tacrolimus. Cyclosporine and tacrolimus have unacceptable interactions with rifamycins.
5. Pulmonary silicosis
6. Central nervous system TB
7. Weight < 40 kg or > 85 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients, by regimen, having negative sputum cultures at completion of eight weeks (40 doses) of treatment | completion of eight weeks (40 doses) of treatment
The proportion of patients, by regimen, who permanently discontinue the assigned study treatment for any reason during the first eight weeks | during the first eight weeks of treatment

SECONDARY OUTCOMES:
time to culture-conversion | 2-, 4-, 6-, and 8-week cultures (10, 20, 30, 40 doses)
proportion of patients with any Grade 3 or 4 adverse reactions | 8 weeks
correlation of the MGIT/BACTEC liquid culture growth index and other mycobacterial and clinical biomarkers with time to culture conversion and treatment failure | duration of TB treatment
compare adverse events and 2-month culture conversion rates among HIV-infected patients vs. HIV-uninfected patients | 8 weeks
• To determine the tolerability and safety, and estimate the antimicrobial activity, of experimental regimens that include higher doses of rifapentine. | 8 weeks.
  • To determine the tolerability and safety, and estimate the antimicrobial activity, of experimental regimens that include isoniazid + pyrazinamide + ethambutol plus either rifapentine 15 mg/kg/dose or rifapentine 20 mg/kg/dose, all administered daily. Assessment of these doses of rifapentine will be performed as an extension to the main study after enrollment in the main study has been completed.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dorman, MD, Principal Investigator — Johns Hopkins University; Neil Schluger, MD, Study Chair — Columbia University; Jason Stout, MD, Study Chair — Duke University
Locations (29):
- United States (23):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of Southern California Medical Center, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California, San Francincisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington DC Veterans Administration Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital, Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - Veterans Administration Tennessee Valley Health Care System, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Veterans Administration Medical Center, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Hopital Universitario Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (2):
  - University of Manitoba, Winnepeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec
- Nelson R Mandela School of Medicine, Durban, KwaZulu-Natal, South Africa
- Agencia de Salut Publica, Barcelona, Spain
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Result] Dorman SE, Goldberg S, Stout JE, Muzanyi G, Johnson JL, Weiner M, Bozeman L, Heilig CM, Feng PJ, Moro R, Narita M, Nahid P, Ray S, Bates E, Haile B, Nuermberger EL, Vernon A, Schluger NW; Tuberculosis Trials Consortium. Substitution of rifapentine for rifampin during intensive phase treatment of pulmonary tuberculosis: study 29 of the tuberculosis trials consortium. J Infect Dis. 2012 Oct 1;206(7):1030-40. doi: 10.1093/infdis/jis461. Epub 2012 Jul 30. PMID 22850121
- [Derived] Gewitz AD, Solans BP, Mac Kenzie WR, Heilig C, Whitworth WC, Johnson JL, Nsubuga P, Dorman S, Weiner M, Savic RM; Tuberculosis Trials Consortium of the Centers for Disease Control and Prevention. Longitudinal Model-Based Biomarker Analysis of Exposure-Response Relationships in Adults with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0179420. doi: 10.1128/AAC.01794-20. Epub 2021 Jul 12. PMID 34252302
- [Derived] Jarsberg LG, Kedia K, Wendler J, Wright AT, Piehowski PD, Gritsenko MA, Shi T, Lewinsohn DM, Sigal GB, Weiner MH, Smith RD, Keane J, Jacobs JM, Nahid P. Nutritional markers and proteome in patients undergoing treatment for pulmonary tuberculosis differ by geographic region. PLoS One. 2021 May 5;16(5):e0250586. doi: 10.1371/journal.pone.0250586. eCollection 2021. PMID 33951066
- [Derived] Weiner M, Gelfond J, Johnson-Pais TL, Engle M, Johnson JL, Whitworth WC, Bliven-Sizemore E, Nsubuga P, Dorman SE, Savic R; Pharmacokinetics/Pharmacodynamics Group of Tuberculosis Trials Consortium. Decreased plasma rifapentine concentrations associated with AADAC single nucleotide polymorphism in adults with tuberculosis. J Antimicrob Chemother. 2021 Feb 11;76(3):582-586. doi: 10.1093/jac/dkaa490. PMID 33374006
- [Derived] Dorman SE, Savic RM, Goldberg S, Stout JE, Schluger N, Muzanyi G, Johnson JL, Nahid P, Hecker EJ, Heilig CM, Bozeman L, Feng PJ, Moro RN, MacKenzie W, Dooley KE, Nuermberger EL, Vernon A, Weiner M; Tuberculosis Trials Consortium. Daily rifapentine for treatment of pulmonary tuberculosis. A randomized, dose-ranging trial. Am J Respir Crit Care Med. 2015 Feb 1;191(3):333-43. doi: 10.1164/rccm.201410-1843OC. PMID 25489785